CLINICAL TRIAL: NCT06800014
Title: Investigation of the Effectiveness of Wearable Activity Trackers and Mobile Application-Supported Telerehabilitation in Individuals With Cerebral Palsy
Brief Title: Effectiveness of Wearable Trackers and Telerehabilitation in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024/02-29
Record Dates: First submitted 2025-01-24; First posted 2025-01-29 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-01

CONDITIONS: Cerebral Palsy (CP); Telerehabilitation; Physical Activity
MeSH Terms: conditions — Cerebral Palsy; Motor Activity | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (Experimental)
  Interventions: Other: Telerehabilitation
- Control (Experimental)
  Interventions: Other: Conventional exercise

INTERVENTIONS:
Other: Telerehabilitation — Participants in the telerehabilitation group will receive weekly home exercise instructions through a mobile application installed on their or their caregivers' smartphones, in addition to their standard rehabilitation program. These instructions will include videos, reminders, and directives for the exercises, with compliance monitored through mini-surveys delivered via the app.
  Arms: Telerehabilitation
Other: Conventional exercise — Participants in the conventional exercise group will continue their standard rehabilitation program supplemented with printed home exercise instructions, including visuals and text, similar to the content provided to the TG.
  Arms: Control

SUMMARY:
The inadequate number of rehabilitation sessions and the difficulties in accessing rehabilitation services for people with cerebral palsy result in delayed progress and low levels of physical activity for these people. As a result, it is well known that daily life often hinders the implementation of prescribed home programmes, leading to neglect. In the rehabilitation of people with cerebral palsy, physiotherapists face difficulties in monitoring patients and ensuring compliance with home exercise programmes. Both people with cerebral palsy and their carers often experience dissatisfaction and lack of motivation regarding the monitoring and control of development and activity.

This study aims to evaluate the effectiveness of a telerehabilitation programme supported by a mobile application and a wearable activity tracker, in addition to a standard rehabilitation programme, on physical activity levels, quality of life, sleep quality, balance, activity participation and motivation, and patient satisfaction in people with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 14 and 18 years old
* Diagnosed with cerebral palsy
* Currently enrolled in a regular rehabilitation programme
* Level 1-3 according to Gross Motor Function Classification System (GMFCS)
* No cognitive impairments affecting the understanding of exercise programmes
* Voluntary informed consent to participate
* No recent surgeries (e.g. botox, muscle relaxation) within the past 6 months
* No socioeconomic issues related to the use of smart devices

Exclusion Criteria:

* The impact of recent surgical procedures or medical interventions on physical performance.
* The influence of health conditions that affect the entire body and physical performance.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-08-07 (Actual)

PRIMARY OUTCOMES:
Physical Activity Questionnaire for Adolescents | Prior to the commencement of the study and following a period of six weeks from the initiation of the application.
  The PAQ-A was developed by Kowalski et al. in 1997 to assess physical activity levels in adolescents (Kowalski et al., 2004). It is suitable for the 14-20 age group. The questionnaire consists of nine questions and assesses physical activity levels over the past seven days. The Turkish validity and reliability study was conducted in 2017. PAQ-A contains eight questions scored between 1 and 5, with a ninth question asking about any condition that might have prevented physical activity during the past week. A score of "1" indicates low-intensity physical activity, while "5" indicates high-intensity physical activity. The ninth question is not included in the scoring. The total score is calculated by averaging the scores of all questions (Aygün Polat, 2017).
Physical Activity Enjoyment Scale | Prior to the commencement of the study and following a period of six weeks from the initiation of the application.
  The PAES is a satisfaction scale developed by Mullen et al., consisting of eight items rated on a 7-point Likert scale (Mullen, 2011). The Turkish validity and reliability study was conducted by Bozkurt et al. (Bozkurt et al., 2022).

SECONDARY OUTCOMES:
Cerebral Palsy Quality of Life Questionnaire for Teen | Prior to the commencement of the study and following a period of six weeks from the initiation of the application.
  The CP-QoL Teen scale is a quality-of-life questionnaire designed for adolescents with cerebral palsy (Davis et al., 2013). Its Turkish adaptation was carried out by Çelik et al. (Çelik, 2012). The CP-QoL Teen scale has two versions: one for caregivers and one self-report version for adolescents. The adolescent self-report version consists of six categories: family and friends, school, participation, communication, health, special equipment, and pain and discomfort. These categories are evaluated under four sections: general well-being and participation, communication and physical health, school situation, and social well-being. The caregiver version includes two additional categories: service assessment and family health (Davis et al., 2013). Scoring involves two steps:
  1. Items are transformed to a scale with a possible range of 0-100;
  2. The algebraic mean of item values is computer for each domain.
Pittsburgh Sleep Quality Index | Prior to the commencement of the study and following a period of six weeks from the initiation of the application.
  The PSQI is a scale that provides information on sleep quality and the type and severity of sleep disorders in the past month (Buysse et al., 1989). Sleep quality is evaluated based on sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleep medication, and daytime dysfunction. The Turkish validity and reliability study of the scale was conducted by Ağargün et al. (Ağargün et al., 1996). Each question is scored between 0 and 3, with higher scores indicating poorer sleep quality. A total score of less than 5 indicates "Good sleep quality," while a score of 5 or above indicates "Poor sleep quality."
Trunk Control Measurement Scale | Prior to the commencement of the study and following a period of six weeks from the initiation of the application.
  The TCMS is a valid and reliable scale for assessing trunk control in individuals with cerebral palsy (Heyrman, 2011). The Turkish validity and reliability study was conducted by Özal et al. (Özal, 2019). The TCMS evaluates two main components of trunk control during functional activities: maintaining balance within the support surface and actively moving body parts. Therefore, the TCMS consists of two main sections: static sitting balance and dynamic sitting balance.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Sciences University, Kütahya, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No